CLINICAL TRIAL: NCT03590444
Title: Treatment of Diabetic Macular Edema (DME) With Intravitreal Anti-vascular Endothelial Growth Factor (Anti-VEGF) and Prompt Versus Deferred Focal Laser During Long-term Follow-up and Identification of Prognostic Retinal Markers
Brief Title: Treatment of Diabetic Macular Edema (DME) With Anti-VEGF and Focal Laser
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Christopher Schütze, Ass.Prof., MD, PhD, Ass.Prof.MD, PhD, Hospital Hietzing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 10-147-0910
Record Dates: First submitted 2018-06-14; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Retinal Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prompt laser group (Active Comparator): Eyes of eligible patients will be randomized (ratio 1:1) and receive ranibizumab and focal/grid laser on the same day (prompt' group, 25 eyes, 50%).
  Interventions: ranibizumab and focal/grid laser on the same day [Ranibizumab (Ranibizumab 0.5 MG/0.05 ML Intraocular Solution]
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution
- Deferred laser group (Active Comparator): Eyes of eligible patients will be randomized (ratio 1:1) and receive ranibizumab and focal/grid laser on one week prior to laser treatment (deferred' group, 25 eyes, 50%).
  Interventions: ranibizumab and focal/grid laser on one week prior to laser treatment [Ranibizumab 0.5 MG/0.05 ML Intraocular Solution]
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution

INTERVENTIONS:
Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution — Focal laser treatment will be performed using argon laser photocoagulation (VISULAS 532s®, Carl Zeiss Meditec) operating at 532nm and Ranibizumab 0.5 MG/0.05 ML Intraocular Solution.
  Ranibizumab 0.5 MG/0.05 ML Intraocular Solution
  Other Names: Focal grid laser

SUMMARY:
Long-term follow-up of patients with diabetic macular edema (DME) treated with intravitreal anti-vascular endothelial growth factor (anti-VEGF) combined focal laser and identification of prognostic morphological characteristics.

DETAILED DESCRIPTION:
Long-term follow-up of patients with diabetic macular edema (DME) treated with intravitreal anti-vascular endothelial growth factor (anti-VEGF) combined focal laser and identification of prognostic morphological characteristics.

Prospective clinical trial (50 treatment-naive eyes) with DME randomized 1:1 receiving intravitreal ranibizumab (0.5 mg/0.05 ml) and prompt grid laser compared to ranibizumab and deferred laser. Morphological characteristics potentially relevant for prognosis were assessed at baseline, month 6, month 9, year 1, 2, 3, 4 and 5 of follow-up.

Grid laser and ranibizumab therapy is expected to be effective in DME management during long-term follow-up. Immediate combined therapy will likely signify a trend of functional superiority in an early disease phase. Intraretinal hyperreflective material in SD-OCT will likely negatively related to BCVA.

ELIGIBILITY:
Inclusion criteria:

* DME that will be detected clinically and on FA as well as on SD-OCT [diffuse macular edema with central retinal thickness (CRT) ≥300µm involving the center of the macular area]
* Patients will be included into the present study following informed consent
* Best-corrected-visual-acuity (BCVA) between 0.06 (1.2logMAR) and 0.63 (0.20logMAR).

Exclusion criteria:

* Eyes with other retinal diseases [i.e. age-related macular degeneration (AMD) and associated choroidal neovascularization (CNV), cystoid macular edema (CME) of other origin (e.g. uveitis, Irvine-Gass syndrome, retinal vein occlusion), or retinal dystrophies]

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Functional alterations will be followed during treatment phase, essential for verification of treatment success. Units: Snellen equivalents

SECONDARY OUTCOMES:
Additional morphological characteristics in spectral Domain SD-OCT | 1 year
  Intraretinal morphological features found in SD- OCT Imaging (i.e. intraretinal morphological changes senn on SD-OCT).
Central retinal thickness | 1 year
  Morphological alterations will be followed during treatment phase, essential for verification of treatment success. Units: Micrometer (retinal thickness)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schütze, Ass.Prof. MD, Principal Investigator — Hietzing Hospital Vienna, Austria
Locations (1):
- Hietzing Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided